CLINICAL TRIAL: NCT07283484
Title: Early Versus Delayed Trial Without Catheter in Men With Acute Urinary Retention: a Randomized Controlled Trial (the RELIEF Study).
Brief Title: Early Versus Delayed Trial Without Catheter in Men With Acute Urinary Retention.
Acronym: RELIEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liselot Ribbert (Other)
Collaborators: Alrijne Hospital (Other); Catharina Ziekenhuis Eindhoven (Other); Canisius Wilhelmina Ziekenhuis (CWZ) (Unknown); Martini Hospital Groningen (Other); Maastricht University Medical Center (Other); Spaarne Gasthuis (Other); St Jansdal Hospital (Other); Ziekenhuisgroep Twente (Other); Zuyderland Medical Centre (Other)
Responsible Party: Sponsor-Investigator, Liselot Ribbert, Study Director, Isala
Organization: Isala (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL-009284; 10390032310057 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2025-11-14; First posted 2025-12-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Urinary Retention; Benign Prostate Obstruction; Benign Prostate Hyperplasia; Benign Prostate Hypertrophy(BPH)
Keywords: RELIEF; Acute Urinary Retention; Urinary Retention; TWOC; Trial Without Catheter; bladder catheter; urinary catheter; catheter removal; catheter withdrawal; Benign prostate obstruction; BPO; Benign prostate hyperplasia; BPH
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Retention

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel-group, non-inferiority trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TWOC after 3 days (Experimental)
  Interventions: Procedure: TWOC after 3 days
- TWOC after 14 days (Active Comparator)
  Interventions: Procedure: TWOC after 14 days

INTERVENTIONS:
Procedure: TWOC after 3 days — A ''trial without catheter'' (TWOC procedure) will be conducted 3 days after catheterization.
  Arms: TWOC after 3 days
Procedure: TWOC after 14 days — A ''trial without catheter'' (TWOC procedure) will be conducted 3 days after catheterization.
  Arms: TWOC after 14 days

SUMMARY:
Acute urinary retention (AUR) is a sudden and painful condition. It occurs when a person is unable to urinate. In men, AUR is most often caused by an enlarged prostate, known as benign prostatic hyperplasia (BPH), which blocks the urethra. The first steps in treatment are to insert a catheter to empty the bladder and to start medication that acts on the prostate (an alpha-blocker). After some time, the catheter is removed during a so-called "Trial Without Catheter" (TWOC) to see whether the patient can urinate normally again.

At present, it is unclear how long a catheter should remain in place before this trial is performed. In Dutch hospitals, the duration varies widely: in some hospitals, the catheter is removed after only a few days, while in others it stays in place for two weeks or longer. A longer catheter duration can cause more discomfort and complications, such as urinary tract infections or blood in the urine. Therefore, it is important to determine whether a shorter catheterization period is equally effective and safe compared to a longer one.

The RELIEF study investigates whether a short catheter duration of three days is as safe and effective as the current average of fourteen days. A total of 478 men with acute urinary retention will participate in this nationwide randomized controlled trial. All participants will receive a catheter and start (or continue) treatment with an alpha-blocker. They will then be randomly assigned to one of two groups: one group will have the catheter removed after three days, and the other group after fourteen days.

The main question is whether a shorter catheter duration is as successful as a longer one. Success means that the patient can urinate normally after catheter removal, without needing to have the catheter replaced. The study will also compare the number of complications, patients' experiences with the catheter, their quality of life, and the overall healthcare costs.

By conducting this study, doctors will gain better evidence on the optimal timing of catheter removal in men with AUR. The goal is to avoid unnecessarily long catheterization, reduce discomfort and complications, and improve the quality of care for men with AUR. The results of the RELIEF study may help improve the management of AUR, making care more consistent, efficient, and patient-friendly both in the Netherlands and abroad.

DETAILED DESCRIPTION:
not aplicable

ELIGIBILITY:
Inclusion Criteria:

* Adult men (≥18 years)
* Diagnosis of acute urinary retention (AUR) treated with a transurethral catheter (TUC) and alpha-blocker therapy (tamsulosin, silodosin, or alfuzosin)
* Mentally competent and able to understand the potential benefits and burdens of study participation
* Provision of written or digital informed consent

Exclusion Criteria:

* Failed prior TWOC within the preceding 30 days
* Initial urinary retention volume >1500 mL
* Neurogenic bladder dysfunction (e.g., multiple sclerosis, spinal cord injury, spina bifida)
* History of prostate cancer with ISUP grade group ≥2
* History of active bladder cancer or ongoing surveillance for bladder cancer
* Urinary retention occurring within 72 hours after surgery (postoperative urinary retention)
* History of lower urinary tract surgery (e.g., bladder augmentation, urethral surgery, or prostate surgery)
* AUR suspected to be caused by bladder stones
* Suspected urethral stricture, clot retention, or urosepsis
* Contraindication to alpha-blocker therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2027-09-04 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Re-catheterization rate after TWOC. | Either 3 or 14 days after catheterization, depending on study group allocation.

SECONDARY OUTCOMES:
Patient reported outcomes - IPSS | Days 3 and 12 after catheter insertion, and at 1, 2, 3, and 6 months.
  Lower urinary tract symptoms measured by the International Prostate Symptom Score (IPSS).
  IPSS is a self-reported score assessing urinary symptoms, including voiding and storage symptoms.
  Range: 0 to 35 (higher scores indicate more severe symptoms).
Patient reported outcomes - EQ-5D-5L | Days 3 and 12 after catheter insertion, and at 1, 2, 3, and 6 months.
  General health-related quality of life measured by the EuroQol 5 Dimensions, 5 Levels questionnaire (EQ-5D-5L) EQ-5D-5L assesses health status across 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Range: 0 to 1 for the index score (higher scores indicate better health); Visual Analogue Scale (VAS) range: 0 to 100 (higher scores indicate better health).
Patient reported outcomes - ICIQ-LTCqol | Days 3 and 12 after catheter insertion, and at 1, 2, 3, and 6 months.
  Catheter-related symptoms and concerns measured by the International Consultation on Incontinence Questionnaire - Long-Term Catheter Quality of Life (ICIQ-LTCQoL) ICIQ-LTCQoL assesses the impact of long-term catheter use on quality of life, including symptoms and concerns.
  Range: 0 to 21 (higher scores indicate more concern and poorer quality of life).
Process related outcomes - Catheter-related complications | Up to 18 months after catheter insertion.
  Catheter related complications (e.g., macroscopic hematuria, CAUTI, urosepsis, catheter related pain or other catheter related problems, urethral strictures), assessed through medical record review and telephone evaluation.
Resource related outcomes - Health care costs | Up to 6 months after catheter insertion (iMCQ assessed at 3 and 6 months).
  Direct health care costs, including costs of (re)catheterization, diagnosis and treatment of complications, and hospital admissions, assessed through medical record review and the iMTA Medical Consumption Questionnaire (iMCQ).
Resource related outcomes - Productivity losses | Up to 6 months after catheter insertion (iPCQ assessed at 1, 2, 3, and 6 months).
  Productivity losses (social costs) assessed using the iMTA Productivity Cost Questionnaire (iPCQ).

CONTACTS AND LOCATIONS:
Overall Officials: Bart P.W. Witte, MD, PhD, Principal Investigator — Isala; Marco H. Blanker, Professor, MD, PhD, Study Chair — University Medical Center Groningen; Liselot L.A. Ribbert, MD, PhD candidate, Study Director — Isala
Locations (11):
- Netherlands (11):
  - St. Jansdal, Harderwijk, Gelderland
  - Canisius Wilhelmina Hospital, Nijmegen, Gelderland
  - Zuyderland Ziekenhuis, Heerlen, Limburg
  - Maastricht University Medical Center+, Maastricht, Limburg
  - Catharina Hospital, Eindhoven, North Brabant
  - OLVG, Amsterdam, North Holland
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - Ziekenhuisgroep Twente, Hengelo, Overijssel
  - Isala, Zwolle, Overijssel
  - Martini Hospital, Groningen, Provincie Groningen
  - Alrijne Hospital, Leiderdorp, South Holland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT07283484/Prot_SAP_000.pdf